CLINICAL TRIAL: NCT06437665
Title: The Tech-wise Driver: Exploring the Sustained Efficacy and Technology Acceptance of Targeted ADAS for Older Drivers
Brief Title: Tech-wise Driver (Technology Acceptance of Targeted ADAS for Older Adults)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Liliana Alvarez Jaramillo, Associate Professor, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R5570A12
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Older Adults; Driving; Simulator
Keywords: Simulator driving, ADAS, Older Adults

STUDY DESIGN:
Intervention Model Description: The parallel model involves comparing two distinct groups, in this case, older drivers (≥65 years of age), who are randomly assigned to either receive ADAS-integrated driver simulation training or driving-simulator training alone. This model allows for a direct comparison between the two groups regarding the effectiveness of the targeted ADAS intervention on driving performance.
Masking Description: Masking, also known as blinding, refers to the practice of concealing information about the intervention assignment from certain parties involved in a study to reduce bias. In the described study, the masking applies to the Outcomes Assessor, who is an independent blinded occupational therapist responsible for evaluating the driving performance of participants. This means that the Outcomes Assessor will not be aware of which group (ADAS-integrated driver simulation training or driving-simulator training alone) each participant belongs to during the assessment process, helping to ensure an unbiased evaluation of the study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADAS-integrated driver simulation training (Experimental): The intervention administered in this study is ADAS-integrated driver simulation training. Participants in this arm will undergo training sessions using a high-fidelity driving simulator equipped with Lane Departure Warning (LDW), Cruise Control (CC), and Forward Proximity Warning (FPW) technologies. These technologies are designed to assist older drivers (≥65 years of age) in improving their driving performance and reducing critical driving errors. The training will simulate real-world driving scenarios to help participants become familiar with and effectively use these ADAS features.
  Interventions: Behavioral: The intervention name in this study is ADAS-integrated driver simulation training.

INTERVENTIONS:
Behavioral: The intervention name in this study is ADAS-integrated driver simulation training. — The intervention involves providing older drivers (≥65 years of age) with training sessions utilizing a high-fidelity driving simulator. This training focuses on the integration and use of Lane Departure Warning (LDW), Cruise Control (CC), and Forward Proximity Warning (FPW) technologies, collectively referred to as ADAS. The training is designed to familiarize participants with these advanced driver assistance systems, enabling them to effectively utilize these features while driving.

SUMMARY:
The tech-wise driver: Exploring the sustained efficacy and technology acceptance of targeted ADAS for older drivers A significant percentage of road traffic fatalities registered in Canada occurred among older adults. According to the studies, the Advanced Driver Assistance Systems (ADAS) can enhance the safety and mitigate the age-related declines of older drivers. Whether sustained use results in declines in driving performance in older drivers relying on ADAS remains largely unexplored. This is problematic given emerging evidence on ADAS use by older drivers. Furthermore, exploring changes in ADAS technology acceptance in relation to sustained use can inform the correlation between perceived safety and intention to use.

The investigators hypothesize that, compared to driving simulator training alone, lane departure warning (LDW), cruise control (CC), and forward proximity warning (FPW) technology will result in a sustained decrease of critical driving errors in this population; and that exposure to the technology will increase participants' perceived usability and ease of use. To achieve this goal, the investigators will explore the determination of sustained efficacy, establish the impact of technology exposure, evaluate the concurrent validity of a computerized model of driving error type and severity using trained occupational therapy in-vehicle evaluation as the criterion, when evaluating older drivers 'performance.

Our findings may significantly impact the ability of older drivers to choose in-vehicle technologies, and our study will be the first to assess the criterion validity of a simulator-derived computerized model against the findings of an evaluator-based functional assessment.

DETAILED DESCRIPTION:
The driving simulator will be used to collect data on drivers in driving scenarios that include situations that may be more challenging for some drivers, e.g., pedestrian stepping into a crosswalk, a vehicle pulling out of a parking spot, a vehicle suddenly changing lanes. Vehicle data and gaze data will be collected for drivers along with images from the simulated environment. The simulator will measure driving performance through metrics generated from the simulator, e.g. pedal (i.e., gas and brake) reaction time, vehicle velocity, headway distance/time, etc.

Participants: Licensed older drivers (≥65 years of age) will be included in this study. Participants will be excluded if they have neurological or psychiatric conditions that would preclude full participation in driving activity, or if they take medications that may have a sustained negative impact on their mental and/or physical functioning during driving.

Sample Size: A sample size of n=68 will be recruited to achieve 80% power to detect a medium effect size of .50 based on a two-sided significance test with a significance level of 0.05.

Procedure:

1. Interested potential participants will reach to the team, using the information distributed during recruitment.
2. Upon confirm eligibility criteria, the first session will be scheduled.
3. Participants will receive a parking pass to park on the premises.
4. The first session will take approximately 1 hr to complete.
5. The objective of the study will be reviewed with each participant and they will be shown the simulator.

2.b. Participants will complete a battery of paper and pencil and computer tests. Of these tests, the first will be vision screening testing to make sure they meet inclusion criteria. Visual acuity (monocular and binocular) will be assessed via Snellen vision charts; visual acuity, peripheral fields, contrast sensitivity, color discrimination, depth perception, lateral phorias and vertical phorias will be assessed via the Optec 5000® Visual Analyzer (Stereo Optical Company, Inc., Chicago, IL). After vision screening, participants will complete an intake form. This is a standardized intake form adapted by the research team which will collect the following information: age, gender, preferred method of contact information for scheduling purposes, self-identified ethnicity, level of education, occupation, and medications. The questions regarding ethnic origin and population group are based on Statistics Canada updated standards.

2.c. Driving History and Habits: The participants will complete several tests germane to their driving history. First, participants will complete a driving history form adapted by the research team (based on Ali et al., 2014). The form will collect information in three sections. Section one will include age at which participants obtained their first license, type of vehicle participants normally drive, whether participants have been involved in a motor vehicle crash and previous use of ADAS technology. Second, participants will complete the computer-based Useful Field of View (UFOV). The UFOV is a standardized test which assesses visual perception and attention (Edwards et al., 2005). This test has shown to be correlated with driving performance among older drivers. The UFOV consists of three subtests that assess attention, divided attention, and selective attention. Finally, the participants will complete the Comprehensive Trail Making Test (CTMT), a normed test in which participants are presented with a standardized set of five visual search and sequencing tasks using pen and paper (Reynolds, 2002).

Rapid Pace Walk Administration: A physical assessment involving walking at a brisk pace, potentially used to evaluate gait and mobility, which can impact a person's ability to operate pedals and controls in a vehicle.

Finger to Nose Administration: A motor coordination test where the participant touches their nose with their finger, assessing fine motor skills and coordination relevant for tasks like steering and operating switches while driving.

Adelaide Self-Efficacy Driving Scale: A self-report questionnaire assessing the participant's confidence and perceived ability in various driving situations, helping to understand their subjective assessment of their driving skills.

Modified Simulator Sickness Questionnaire: A questionnaire measuring symptoms of simulator sickness or discomfort experienced during driving simulation sessions, important for evaluating the usability and comfort of simulation-based assessments.

Driving Simulation Evaluation Form: A structured form or checklist used to evaluate the participant's performance and behavior during driving simulation scenarios, providing objective data on driving skills and behaviors.

Manchester Driving Behavior Questionnaire: A questionnaire assessing self-reported driving behaviors and attitudes, offering insights into the participant's driving style, risk perception, and adherence to traffic rules.

The post-assessment tests generally involve reassessing specific aspects measured during the baseline assessment or evaluating any changes or improvements following interventions or training.

2.d. Following these tests, participants will complete their simulation drives. The investigators will employ a clinical driving simulator (DriveSafety Inc., Salt Lake City, UT). Prior to each drive, participants will be exposed to an acclimation drive. Acclimation drives are part of a mitigation protocol aimed at reducing the likelihood of participants experiencing discomfort caused by simulation. Such drives last no longer than 7 minutes, and slowly introduce the participant to the simulation, starting with simple maneuvers (e.g., accelerate ad stop) and progressively introducing more complex maneuvers (e.g. turning).

2.e. Each Participants will then complete a randomized 15-minute drive. Participants will then take part in three sets of four training sessions in which the ADAS will be simulated (experimental group) or a training script will be provided (control). After each set of four drives, a simulator assessment post-test will be completed with the final post-test also including the battery of clinical assessments. Available routes will be randomly allocated and counterbalanced across participants. All drives will be recorded (frontal view of the driver as well as simulated drive). Once a participant has completed all drives, the recordings will be sent to a blinded trained evaluator (occupational therapist and driving rehabilitation specialist). The study will use a high-fidelity clinical driving simulator (DriveSafety Inc) configured with three 19 inch flat-panel displays; 110-degree field of view; 1920 x 1080 pixels/screen. Raw files will be used to develop and compute the model for comparison. The drive using the simulator will be recorded (mp4). This will allow the post-drive evaluation of the number and type of driving errors conducted by the research team. In addition to recording the simulation drive, a camera located in the simulator records the face of the driver to enable scoring of visual scanning errors. All video files are stored in the password protected research drive connected to the simulator computer in the research lab, and only accessible to members of this research team. There will also be a stereo camera attached to the simulator for collecting gaze information of the driver. This camera is connected to a computer running gaze analysis software and records only the gaze directions (as vector in the 3D space of the camera) and head direction (also a vector in the 3D space of the camera). This data is numeric and will be stored using the identifier assigned to the participant; no images are collected from this camera. Prior to and after each drive, the Adapted Motion Sickness Questionnaire will be used to monitor for any signs of simulator sickness. If a participant scores over 5 in any of the items, the session will be suspended, the participants remunerated and provided with access to water, ginger ale, crackers, and cool room. No further drives will be attempted to avoid any risk of increasing simulator sickness.

2.f. After the driving session, the research team will thank the participant and provide remuneration.

3.In order to give the team access to the driving simulator metrics of each drive, a password protected One Drive folder within Western's license will be used. Only deidentified driving simulator data will be uploaded to the One Drive.

ELIGIBILITY:
Inclusion Criteria:

* Must be 65 years of age or older.
* Must hold a valid driver's license.

Exclusion Criteria:

* Neurological or psychiatric conditions that would preclude driving
* Use of psychotropic medications that may have a sustained negative impact on mental and/or physical functioning

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of driving errors | The study will span over a 12-week period, encompassing pre-test, post-test 1, and post-test 2 assessments.
  This outcome aims to assess the sustained efficacy of a targeted Advanced Driver Assistance Systems (ADAS) intervention comprising Lane Departure Warning (LDW), Cruise Control (CC), and Forward Proximity Warning (FPW) technologies on the driving performance of older drivers (≥65 years). The study compares the performance of participants who receive ADAS-integrated driver simulation training against those who undergo driving-simulator training alone. The primary focus is on measuring the decrease in critical driving errors, as evaluated by an independent blinded occupational therapist, across post-test intervals.
Type of driving errors | The study will span over a 12-week period, encompassing pre-test, post-test 1, and post-test 2 assessments.
  The blinded evaluator will record type pf driving errors, to establish if there is a decrease in the number of critical driving errors (i.e. those requiring physical intervention from an instructor).

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Alvarez, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Western University, London, Ontario, Canada